CLINICAL TRIAL: NCT03138876
Title: EEG Cap Placement for Expedited Identification of Non-Convulsive Status Epilepticus
Brief Title: EEG Cap for Identification of Non-Convulsive Status Epilepticus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, William Tatum, DO, Professor of Neurology, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 16-008778
Record Dates: First submitted 2017-05-01; First posted 2017-05-03 (Actual); Results first posted 2019-10-25 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Nonconvulsive Status Epilepticus; Subclinical Seizure; Altered Mental Status; Nonepileptic Seizures; Encephalopathy
MeSH Terms: conditions — Status Epilepticus; Epilepsies, Partial; Seizures; Brain Diseases

STUDY DESIGN:
Intervention Model Description: Subjects may be treated for NCSE based on EEG cap findings, but only following standard practice. The study is designed to identify NCSE, not to assess treatment of NCSE.
Masking Description: There will be blinded EEG assessment in terms of the EEG readers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- EEG Cap (Other): Single arm study, where every participant gets assessed by EEG cap and then standard EEG. Some subjects may be treated with anti-seizure medications before standard EEG, due to ethical responsibility, if clear NCSE is identified on cap EEG. If the subject is treated with anti-seizure medication, the primary care provider will choose which medication will be given.
  Interventions: Device: EEG Cap; Drug: Anti-seizure medication; Procedure: Standard EEG

INTERVENTIONS:
Device: EEG Cap — Patient will be fitted with an EEG cap by the on-call neurology resident to assess for NCSE.
  Other Names: Electro-Cap
Drug: Anti-seizure medication — Patients may be treated for NCSE or seizures based on EEG cap findings, if the findings are clear to an attending EEG reviewer. If the subject is treated with anti-seizure medication, the primary care provider will choose which medication will be given.
Procedure: Standard EEG — An electroencephalogram (EEG) is a test used to find problems related to electrical activity of the brain. An EEG tracks and records brain wave patterns. Small metal discs with thin wires (electrodes) are placed on the scalp, and then send signals to a computer to record the results.

SUMMARY:
Altered mental status (AMS) is one of the most common reasons for inpatient neurology consultation. Non-convulsive status epilepticus (NCSE) is frequently on the differential diagnosis of the patient with AMS. NCSE becomes more refractory to treatment after one hour of seizure activity, making rapid identification and treatment of NCSE of great clinical importance. Currently, an electroencephalogram (EEG) technologist must be called in from home during non-workday hours in order to obtain a stat EEG. The investigators propose the time required for diagnosis of NCSE at Mayo Clinic can be significantly decreased with rapid placement of an EEG cap by the onsite neurology residents.

DETAILED DESCRIPTION:
At the completion of neurology evaluation, if NCSE is in the differential diagnosis according to institution best practice, then consented participants will undergo placement of a large size, 20-channel EEG cap from Electro-Cap International with a Natus E-2-2520-26 electrode board adapter with initiation of recording. The placement of the EEG cap will be restricted to residents formally trained in its placement by an EEG tech. This study will only be performed during times when EEG techs are not available onsite for rapid placement of standard 21-channel EEG electrodes, such as during night-call shifts.

Prior to placement of EEG cap, evaluating staff member will request immediate standard-electrode EEG. The investigators will record time from neurology consultation request to placement of EEG cap as well as time from consultation request to obtaining a standard EEG. The investigators will also record time to confirmation or exclusion of NCSE. Initial diagnosis or exclusion of NCSE will be performed by on call resident, if the resident received prior training regarding EEG cap placement, and attending. Secondary quality assessment will be performed by two independent EEG interpreters blinded to clinical history. Secondary assessment will be qualified as acceptable or inacceptable interpretation based on whether greater or less than 50% of the recording is judged interpretable. Secondary assessment will also include interpretation of NCSE by a third independent reader if there is disagreement between first two. The number of patients excluded from the study will also be recorded, including the reason for exclusion.

ELIGIBILITY:
Inclusion criteria:

1. Patients with suspected NCSE in the Mayo Clinic Florida hospital, emergency room or intensive care unit.
2. Age: Patients of 18 years or older will be included in this study
3. Education: All education levels will be included

Exclusion criteria:

1. Patients younger than 18 years of age.
2. Patients with open head trauma.
3. Patients with anatomy that would preclude EEG cap placement.
4. Patients excluded for anatomical or age-related reasons will be tracked to determine applicability of the EEG cap to the patient population at Mayo Clinic.
5. Pregnant females
6. Large head size not amenable to cap placement
7. Scalp infection
8. Inability to obtain informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2018-08-16 (Actual); Study Completion 2018-08-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Tatum, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferlisi M, Shorvon S. The outcome of therapies in refractory and super-refractory convulsive status epilepticus and recommendations for therapy. Brain. 2012 Aug;135(Pt 8):2314-28. doi: 10.1093/brain/aws091. Epub 2012 May 9. PMID 22577217

RESULTS

PARTICIPANT FLOW:
Groups:
- EEG Cap: Single arm study, where every participant gets assessed by an electroencephalogram (EEG) cap and then standard EEG. Some subjects may be treated with anti-seizure medications before standard EEG, due to ethical responsibility, if clear Non-convulsive status epilepticus (NCSE) is identified on cap EEG. If the subject is treated with anti-seizure medication, the primary care provider will choose which medication will be given.
Period: Overall Study
Arm/Group | EEG Cap
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- EEG Cap: Single arm study, where every participant gets assessed by an electroencephalogram (EEG) cap and then standard EEG. Some subjects may be treated with anti-seizure medications before standard EEG, due to ethical responsibility, if clear NCSE is identified on cap EEG. If the subject is treated with anti-seizure medication, the primary care provider will choose which medication will be given.
Arm/Group | EEG Cap
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (18.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Time Difference Between EEG Cap and Standard EEG Results Reporting
Description: The difference between EEG Cap results reporting time compared to Standard EEG results reporting time measured in minutes.
Time Frame: EEG order through 20 minutes of EEG recording time
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | EEG Cap
Number analyzed (Participants) | 12
minutes | 103.4 (42.6)
Statistical Analysis 1: Comparison: EEG Cap; Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Percentage of Participants Whose EEG Cap Recordings Were Interpretable
Description: The recording will be qualified as acceptable interpretation if greater than 50% of the recording is judged interpretable by board certified electroencephalographers.
Time Frame: approximately 15 minutes after completion of test
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Cap
Number analyzed (Participants) | 20
Participants | 14

3. Secondary Outcome: Number of Subjects Diagnosed With NCSE
Description: The number of subjects with suspected NCSE subsequently confirmed with NCSE after standard EEG.
Time Frame: approximately within 15 minutes after completion of test
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Cap
Number analyzed (Participants) | 20
Participants | 3

4. Secondary Outcome: Number of Subjects for Which the EEG Cap and Standard EEG Results Are in Agreement for the Diagnosis of NCSE
Description: Concordance between cap and standard-electrode diagnostic assessments
Time Frame: approximately 24 hours after completion of both tests
Measure: Count of Participants; unit: Participants
Arm/Group | EEG Cap
Number analyzed (Participants) | 20
Participants | 3

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the EEG testing each subject, over a study period of 11 months.
Arm/Group | EEG Cap
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20
Other Adverse Events (participants affected / at risk) | 0/20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03138876/Prot_SAP_000.pdf